CLINICAL TRIAL: NCT00071019
Title: Dietary Fatty Acids, PPAR Activated Genes, and CHD
Status: Completed | Type: Observational
Sponsor: Harvard School of Public Health (HSPH) (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Hannia Campos, Senior Lecturer, Harvard School of Public Health (HSPH)
Other Study IDs: 1235; R01HL071888 (NIH)
Record Dates: First submitted 2003-10-09; First posted 2003-10-13 (Estimated); Last update posted 2017-04-20 (Actual); Status verified 2017-04

CONDITIONS: Coronary Disease; Cardiovascular Diseases; Heart Diseases; Myocardial Infarction
MeSH Terms: conditions — Coronary Disease; Cardiovascular Diseases; Heart Diseases; Myocardial Infarction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To examine the relationship between genetic and dietary factors that modify the risk of coronary heart disease (CHD).

DETAILED DESCRIPTION:
BACKGROUND:

Coronary heart disease (CHD) is the major cause of death in most industrialized and developing countries. Links between genetic and dietary factors that modify the risk of CHD should give fundamental insight into its causes and improve population-based CHD prevention strategies.

DESIGN NARRATIVE:

The study will identify genes that modulate the association between dietary fatty acids (FAs) and myocardial infarction (MI). The study uses DNA samples obtained during a population-based, case-control study in Costa Rica of 2,150 subjects who experienced myocardial infarctions and 2,150 matched controls. Biochemical measurements, dietary data, and general information are available for this population. One unique aspect of the study is that adipose tissue biomarkers of polyunsaturated FAs will be used to evaluate dietary exposure variables. Adipose tissue biomarkers (i.e., alpha-linolenic and linoleic acid) are very good indicators of intake in this population. Furthermore, this study showed that increased levels of these biomarkers in adipose tissue are strongly associated with decreased risk of MI, whereas an increase in 18:2 trans FAs increase the risk of MI. Gene-diet association studies and a "candidate pathway" approach will be used to elucidate genetic mechanisms that link risk of MI with exposure to polyunsaturated FAs [including cis and trans isomers of linoleic acid (n-6), and alpha-linolenic acid (n-3)]. The focus will be on peroxisome proliferator-activated receptor (PPAR) genes, and PPAR-regulated genes, that are involved in vascular inflammation. Among controls, the investigators will examine whether genetic and dietary factors independently affect biochemical markers (phenotypes) of the proposed genes. They will also test whether these phenotypes are more clearly identified when genetic and dietary factors are examined together. Because polyunsaturated FAs are important as activators of PPARs and their capacity to regulate gene expression at the level of transcription, this metabolic system is a suitable candidate for the study.

ELIGIBILITY:
First acute MI Living in catchment area Randomly selected controls Matched for age sex and area of residence

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hispanic American of mestizo background living in Costa Rica
Sampling Method: Probability Sample
Enrollment: 4547 (Actual)
Dates: Start 2003-09; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hannia Campos, Principal Investigator — Harvard School of Public Health (HSPH)

IPD SHARING:
Plan to Share IPD: No